CLINICAL TRIAL: NCT04881201
Title: Metabolomic Exploration of Dysregulated Lipid Metabolism in MFN2-related CMT2A (CMT2A) Linked to Mitofusin 2
Brief Title: Metabolomic Exploration of Dysregulated Lipid Metabolism in MFN2-related CMT2A (MetaDLM_CMT2A)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A00834-34
Record Dates: First submitted 2021-04-27; First posted 2021-05-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Charcot-Marie-Tooth Disease Type 2A
MeSH Terms: conditions — Charcot-Marie-Tooth disease, Type 2A | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients Charcot-Marie-Tooth (Other)
  Interventions: Procedure: blood sample
- Control subjects (Other)
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — blood sample

SUMMARY:
Charcot-Marie-Tooth (CMT) disease is the commonest sensitivo-motor inherited peripheral neuropathies with a prevalence of about 10-30 per 100,000. To date, more than 80 genes have been found responsible for CMT. Some of these genes code for mitochondrial proteins such as mitofusin 2 (MFN2).

In the last few years, our laboratory has developed strong expertise in metabolomics. The MetaDLM_CMT2A project proposes to produce metabolomic and lipidomic maps in CMT2A plasma from a cohort of genetically and clinically characterized patients with a national recruitment.

In the perspective of future clinical trials, these biomarkers and the better understanding of lipid metabolism defects in CMT2A would be of major interest in monitoring the evolution of the disease and developing specific therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

For all participants :

* Adult person
* Person on an empty stomach at the time of inclusion
* Person who signed the study participation consent form
* Person affiliated or beneficiary of a social security scheme

Patients Charcot-Marie-Tooth :

* Patient with symptoms of Charcot-Marie-Tooth disease on clinical examination clinical examination
* Patient with axonal neuropathy confirmed by an electrophysiological study electrophysiological study with a median nerve conduction velocity > 38 m / s
* Patient with documented pathogenic mutation (class 4 or class 5) in the MFN2 or patient with a variant of uncertain significance, as determined by the laboratory performing the test, if the variant of unknown significance has been found in found in multiple affected individuals in a family and not found in unaffected family members in unaffected family members.

Control subject :

* Each control is matched in age and sex to a case previously included in the study.

Exclusion Criteria:

For all participants :

* Pregnant, breastfeeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person subject to forced psychiatric care
* Person subject to a legal protection measure
* Person unable to give consent

Patients Charcot-Marie-Tooth :

* Patient with a neuropathy other than CMT2A (such as diabetic neuropathy or any other cause of acquired neuropathy) neuropathy or any other cause of acquired neuropathy), medical history of kidney stones kidney stones or cardiovascular risk factors (dyslipidaemia diabetes, severe obesity (BMI >35 kg/m²))
* Patient treated with Idebenone at the time of inclusion. (It is possible to include a patient treated with Idebenone if the treatment was interrupted at least 5 days before)

Control subject :

* Person with neuropathy, medical history of kidney stones or cardiovascular risk factors cardiovascular risk factors (dyslipidaemia, diabetes, severe obesity (BMI >35 kg/m²))

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Compare the metabolomics and lipidomics of CMT2A patients compared to witnesses using high resolution mass spectrometry | at enrollment
  We will compare the metabolomics and lipidomics of CMT2A patients compared to controls using high resolution mass spectrometry, by comparing the presence or not of the metabolites sought thanks to thetechnology developed by the company Biocrates (MxP-Quant-500 kit), allowing testing of 630 polar and lipid metabolites, under conditions close to medical biology.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Angers, maine et loire, France

IPD SHARING:
Plan to Share IPD: No